CLINICAL TRIAL: NCT05457374
Title: A Clinical Study of Portal Vein Embolization and Liver Venous Deprivation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LLX-002
Record Dates: First submitted 2022-07-10; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-05

CONDITIONS: Liver Venous Deprivation

STUDY DESIGN:
Intervention Model Description: Partial hepatectomy+PVE Partial hepatectomy+LVD
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial hepatectomy+LVD (Experimental)
  Interventions: Procedure: LVD
- Partial hepatectomy+PVE (Experimental)
  Interventions: Procedure: PVE

INTERVENTIONS:
Procedure: PVE — Portal vein embolization (PVE) mainly embolizes the portal vein of the resected liver lobe, causing the non-tumor lobe to proliferate, and after tumor lobectomy, the volume of the non-tumor lobe proliferates so that patients with hepatocellular carcinoma that could not be directly surgically resected are given the opportunity to be surgically resected
  Arms: Partial hepatectomy+PVE
Procedure: LVD — Combining PVE and Hepatic Vein Embolization (HVE) in the same procedure
  Arms: Partial hepatectomy+LVD

SUMMARY:
The main obstacle to achieving R0 resection in future liver remnant（FLR） deficient liver cancer is the inability to retain sufficient FLR to avoid postoperative liver failure. From the initial portal vein embolization(PVE), to the later ALPPS, this problem has been solved to some extent. However, both have their own shortcomings. The effect of liver hyperplasia after PVE is poor and the waiting time is long. The incidence of complication and mortality after ALPPS is always the focus of controversy. In recent years, LVD has emerged, combining PVE and HVE in the one operation. This topic will conduct a clinical controlled study of PVE and LVD.

ELIGIBILITY:
Inclusion Criteria:

* ① Age 18 to 75 years old, male or female.

  * hepatocellular liver cancer diagnosed by pathological histology, immunohistochemistry or imaging examination, with large tumor size that cannot be removed in one stage surgery

    * No distant metastasis of the lesion.

      * FLR<20% in patients with normal liver function; FLR<30% in patients with combined fatty liver and receiving chemotherapy; FLR<40% in compensated cirrhosis ⑤ Normal function of major organs other than liver-related functions. ⑥ Subjects voluntarily enrolled in this study, signed informed consent, good compliance, and cooperated with follow-up.

        * Patients who the investigator believes can benefit.

Exclusion Criteria:

* Withdrawal of consent by the subject.

  * Having adverse reactions. ③ Failure to receive treatment due to progression.

    * Death of the patient.

      * Loss to follow-up. ⑥ Others.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
FLR growth rate | 15days
  FLR growth rate between two surgeries

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui province hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No